CLINICAL TRIAL: NCT06293729
Title: A Clinical Study for the Safety and Efficacy of Intravenous Infusion of NGGT006 in Treatment of Refractory Hypercholesterolemia
Brief Title: Safety and Efficacy Study of NGGT006 in Refractory Hypercholesterolemia Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Suzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, Yan Chen, President of Suzhou Municipal Hospital, Suzhou Municipal Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGGT006-P-2302
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Refractory Hypercholesterolemia; Familial Hypercholesterolemia
Keywords: Gene therapy; Low-density lipoprotein cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGGT006 (Experimental): 3 doses of NGGT006 will be administered according to the principle of dose escalation
  Interventions: Drug: NGGT006

INTERVENTIONS:
Drug: NGGT006 — Single intravenous infusion of NGGT006 at low dose (7.5e12vg/kg), medium dose (1.5e13vg/kg) and high dose (3e13vg/kg).

SUMMARY:
This is an early phase 1, open-label, single-center, dose-escalation pilot trial to evaluate the safety and efficacy of an intravenous infusion of NGGT006 in patients with refractory Hypercholesterolemia diagnosed by gene testing for familial hypercholesterolemia. NGGT006 uses adeno-associated virus (AAV) as a vector, carrying a liver specific promoter and codon optimized human LDLR gene, driving the expression of LDLR protein with normal function and promoting the clearance of low-density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
Familial Hypercholesterolemia caused by common genetic mutations can be divided into heterozygous hypercholesterolemia (HeFH, Heterozygous Familial Hypercholesterolemia) and homozygous hypercholesterolemia (HoFH, Homozygous Familial Hypercholesterolemia). Refractory hypercholesterolemia was defined as an LDL-C level of 70 mg/dL or greater, or 100 mg/dL or greater, for patients with or without clinical ASCVD, respectively. A large proportion of patients with familial hypercholesterolemia belong to refractory hypercholesterolemia. This is an early phase 1, open-label, single-center, dose-escalation pilot trial to evaluate the safety and efficacy of a single intravenous infusion of NGGT006 in patients with refractory Hypercholesterolemia diagnosed by gene testing for familial hypercholesterolemia. 3-9 subjects will be enrolled and divided into 3 groups according to the principle of dose escalation, respectively administered intravenous infusion of NGGT006 at low dose (7.5e12vg/kg), medium dose (1.5e13vg/kg) and high dose (3e13vg/kg). All subjects will undergo 52 weeks of treatment observation and further 260 weeks of long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 55 years old;
2. A patient with a clear diagnosis of refractory hypercholesterolemia and confirmed by genetic testing to be familial hypercholesterolemia;
3. AAV binding antibody titer ≤1:80 and AAV neutralizing antibody ≤1:5;
4. 18≤BMI (body mass index)≤35;
5. During the screening period, the subjects have received stable maximum tolerated dose of lipid-lowering drug treatment, but LDL-C was still ≥70mg/dL with clinical atherosclerotic cardiovascular disease; or LDL-C level was ≥ 100 mg/dL without clinical atherosclerotic cardiovascular disease: the highest tolerated dose refers to (the following must be met at the same time):

   ① Moderate to high doses of statins for ≥4 weeks, whether used alone or in combination with other lipid-lowering drugs; exceptions: subjects cannot tolerate statins; or subjects cannot receive statin treatment due to other reasons, such as low BMI, etc.;

   ② Ezetimibe ≥ 4 weeks;

   ③ Alirocumab 150mg Q2W or 300mg Q4W; evolocumab 140mg Q2W or 420mg Q4W; ≥8 weeks; And during the clinical trial process, any adjustment involving the type and dosage of lipid-lowering drugs must be approved by the researcher;
6. Stable healthy diet for ≥12 weeks, and can adhere to a healthy diet throughout the entire clinical trial;
7. Voluntarily sign the informed consent form and be willing to comply with the trial visit plan;
8. Willing to maintain a similar amount and intensity of exercise during the study period as during the baseline period;
9. Maintain good living habits, have no history of alcoholism or alcohol dependence (ICD-10 diagnosis is F10)
10. No new or recurring cardiovascular events (myocardial infarction, cerebral infarction, etc.) within half a year;
11. No stent implantation plan within three months;
12. Female subjects have not had sexual intercourse for 14 days before administration, and their blood tests indicate that they are not pregnant;
13. Subjects of childbearing age agree to use highly effective contraceptive measures for at least 365 days from the time of NGGT006 administration.

Exclusion Criteria:

1. Secondary hyperlipidemia;
2. Use of other drugs or nutritional products that may affect blood lipids (such as fibrates) within 6 weeks;
3. Have received low-density lipoprotein apheresis (LDL apheresis) within the past 2 months;
4. Large weight fluctuations (≥5kg) in the past 2 months;
5. Positive for hepatitis B surface antigen, hepatitis C, human immunodeficiency virus (HIV)，syphilis test or other infections (such as Epstein-Barr virus, Mycoplasma pneumoniae, tuberculosis virus, HPV, Chlamydia pneumoniae, respiratory syncytial virus, Adenovirus and coxsackievirus group B, etc.);
6. Clinically significant abnormalities in liver function test: alanine aminotransferase (ALT) >2 × upper limit of normal (ULN) and/or aspartate aminotransferase (AST) >2 × ULN;
7. RR at the baseline >160/100mmHg (one repeated measurement is allowed);
8. Uncontrollable myocardial infarction or heart failure, and those planning surgery within one year; or new acute coronary syndrome in the past six months;
9. Diabetes diagnosed within 3 months or with poor control (HbA1c >9%);
10. Abnormal thyroid function, or those using thyroid hormone replacement therapy but poorly controlled (TSH within the normal range for <12 weeks);
11. Acute or chronic renal insufficiency;
12. Hemoglobin (Hb) < 120g/L (male), Hb < 110 (female);
13. Abnormal platelet counts or morphology;
14. History or laboratory tests suggestive of thrombosis;
15. Had contraindications to glucocorticoid (e.g., epilepsy, severe schizophrenia, active peptic ulcer)；
16. Used systemic glucocorticoid treatment within 6 weeks before enrollment;
17. Life expectancy less than 1 year;
18. Suffering from malignant tumors such as liver cancer; liver fibrosis;
19. Previous gene therapy treatment;
20. Hypersensitivity to AAV preparations (for example trehalose) or cortisone or immunosuppressants (sirolimus, rituximab, tacrolimus);
21. Suffering from immunodeficiency disease
22. Participation in any other clinical trial within 3 months;
23. Breastfeeding females;
24. Any other condition that may not be appropriate for the study in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (AE) and serious adverse events (SAE) | 52 weeks
  Incidence of AE and SAE, as assessed by physical examinations, clinical laboratory parameters and adverse event reporting
Absolute change and percent change in LDL-C | 52 weeks
  Change in LDL-C concentration from baseline to week 52

SECONDARY OUTCOMES:
Absolute change and percent change in non-high density lipoprotein cholesterol | 52 weeks
  Change in non-HDL-C from baseline to week 52
Absolute change and percent change in apolipoprotein B | 52 weeks
  Change in ApoB from baseline to week 52
Absolute change and percent change in total cholesterol | 52 weeks
  Change in TC from baseline to week 52
Absolute change and percent change in HDL-C | 52 weeks
  Change in HDL-C from baseline to week 52
Absolute change and percent change in triglycerides | 52 weeks
  Change in TG from baseline to week 52
Absolute change and percent change in very low-density lipoprotein cholesterol | 52 weeks
  Change in VLDL from baseline to week 52
Absolute change and percent change in lipoprotein(a) | 52 weeks
  Change in Lp(a) from baseline to week 52
Absolute change and percent change in apolipoprotein A-I | 52 weeks
  Change in apo A-I from baseline to week 52

IPD SHARING:
Plan to Share IPD: No